CLINICAL TRIAL: NCT04881630
Title: Mobile Contingency Management for Smoking Cessation Among Socioeconomically Disadvantaged Adults
Brief Title: Mobile Contingency Management for Smoking Cessation
Acronym: P3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH); M.D. Anderson Cancer Center (Other); University of Florida (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12881; R01CA251451 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-05-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Financial Incentives; Socioeconomic Status; Contingency Management; Mobile Health
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (SC) (Active Comparator): Participants randomized to Standard Care will be offered weekly smoking cessation counseling and pharmacotherapy.
  Interventions: Other: Standard Care (SC)
- Contingency Management (CM) (Experimental): CM participants will receive standard care in addition to small financial incentives for biochemically-verified abstinence.
  Interventions: Behavioral: Automated Mobile Contingency Management (CM); Other: Standard Care (SC)

INTERVENTIONS:
Behavioral: Automated Mobile Contingency Management (CM) — Financial incentives contingent upon smoking abstinence
  Arms: Contingency Management (CM)
Other: Standard Care (SC) — Tobacco cessation telephone counseling and combination nicotine replacement therapy (nicotine patches + nicotine gum/lozenges)

SUMMARY:
The purpose of the proposed project is to evaluate an automated mobile phone-based CM approach that will allow socioeconomically disadvantaged individuals to remotely benefit from financial incentives for smoking cessation. The investigators have previously combined technologies including 1) portable carbon monoxide monitors that connect with mobile phones to remotely verify smoking abstinence, 2) facial recognition software to confirm participant identity during breath sample submissions, and 3) remote delivery of incentives automatically triggered by biochemical confirmation of self-reported abstinence. This automated CM approach will be evaluated in a randomized controlled trial that includes 532 socioeconomically disadvantaged males and females seeking smoking cessation treatment. Participants will be randomly assigned to either telephone counseling and nicotine replacement therapy (standard care [SC]) or SC plus a mobile financial incentives intervention (CM) for biochemically-confirmed abstinence. Participants will be followed for 26 weeks after a scheduled quit attempt. Biochemically-verified 7-day point prevalence abstinence at 26 weeks post-quit will be the primary outcome variable. Cost-effectiveness will be evaluated to inform policy-related decisions. Potential mobile CM treatment mechanisms, including self-efficacy, motivation, and treatment engagement, will be explored to optimize future versions of the intervention.

DETAILED DESCRIPTION:
The primary purpose of the proposed project is to evaluate an automated smartphone-based CM approach that will allow socioeconomically disadvantaged adults to earn financial incentives for smoking cessation without requiring in-person attendance for abstinence verification. The investigators have combined technologies: 1) low-cost carbon monoxide monitors that connect with mobile phones to remotely verify smoking abstinence, 2) facial recognition software to verify the identity of participants while they provide a breath sample, and 3) remote and automated delivery of incentives to a credit card triggered by biochemical confirmation of self-reported smoking abstinence. This CM approach will be evaluated in a randomized controlled trial of 532 socioeconomically disadvantaged males and females seeking smoking cessation treatment. Participants will be randomly assigned to telephone counseling plus nicotine replacement therapy (standard care [SC]) or SC plus a 12-week smartphone-based financial incentives intervention (CM). Participants will be followed for 26 weeks after a scheduled quit attempt, which is 14 weeks after incentives have ended. Cost-effectiveness will be evaluated to inform policy and health care decisions. Potential CM treatment mechanisms, including self-efficacy, motivation, and treatment engagement will be identified to optimize future versions of the intervention. The specific aims are: 1) to evaluate the impact of an automated, mobile phone-based CM approach relative to SC on smoking cessation among socioeconomically disadvantaged adults, 2) to compare the cost-effectiveness of two smoking cessation interventions (CM vs. SC), and 3) to identify mobile CM treatment mechanisms such as motivation to quit, self-efficacy for quitting, and treatment engagement/adherence. The proposed study will evaluate an intervention approach that increases the reach of a potentially effective and cost-effective smoking cessation intervention for socioeconomically disadvantaged smokers. This proposed study is also going to be conducting recruitment nationwide.

ELIGIBILITY:
Inclusion Criteria:

1. report an annual household income of <200% of the federal poverty threshold (i.e., low-income)
2. earn a score ≥4 on the REALM indicating >6th grade English literacy level (i.e., a 7th grade reading level is necessary to complete assessments)
3. are willing to quit smoking 7-14 days after enrollment
4. are ≥ 18 years of age
5. currently smoke ≥ 5 cigarettes per day
6. have a CO level of >6 ppm
7. are willing to abstain from smoking cannabis and other combustible tobacco products (they raise CO levels and mask cigarette abstinence)
8. have no contraindications for NRT
9. Provide a copy/photo of driver's license or other documentation as proof of identity and U.S. residence

Exclusion Criteria

1) do not meet the specified inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Carbon monoxide-verified smoking abstinence | 26 weeks post-quit-date
  The primary outcome measure is carbon monoxide-verified 7-day point prevalence abstinence at 26 weeks post-quit.

SECONDARY OUTCOMES:
Cost-effectiveness | 26 weeks post-quit-date
  The incremental cost effectiveness ratio (ICER) calculated as the difference in mean costs between the new (CM) and standard treatment (SC) divided by the difference in mean effectiveness between the two, estimates additional resources needed to achieve an increase of one unit of effectiveness. The ICER is then compared with published threshold values for cost-effective interventions. The cost model will include all necessary personnel, hardware, and material costs.
Carbon monoxide-verified smoking abstinence | 12 week post-quit-date
  Carbon monoxide-verified 7-day point prevalence abstinence at 12 weeks post-quit-date.
Carbon monoxide-verified smoking abstinence | 8 weeks post-quit-date
  Carbon monoxide-verified 7-day point prevalence abstinence at 8 weeks post-quit-date.
Carbon monoxide-verified smoking abstinence | 4 weeks post-quit-date
  Carbon monoxide-verified 7-day point prevalence abstinence at 4 weeks post-quit-date.
Carbon monoxide-verified smoking abstinence | 26 weeks post-quit-date
  Carbon monoxide-verified 30-day point prevalence abstinence at 26 weeks post-quit-date.

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to investigators upon request, after publication of the primary study findings, and with a data-sharing agreement that specifies the investigator(s) will 1) use the data only for research purposes and not to identify any individual participant, 2) store the data on a secure device (e.g., encrypted, password-protected), and 3) destroy or return the data after completion of the analyses.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be made available to investigators upon request after publication of the primary study findings.
Access Criteria: Data sharing agreement

REFERENCES:
- [Background] Kendzor DE, Businelle MS, Vidrine DJ, Frank-Pearce SG, Shih YT, Dallery J, Alexander AC, Boozary LK, Waring JJC, Ehlke SJ. Mobile contingency management for smoking cessation among socioeconomically disadvantaged adults: Protocol for a randomized trial. Contemp Clin Trials. 2022 Mar;114:106701. doi: 10.1016/j.cct.2022.106701. Epub 2022 Jan 31. PMID 35114409